CLINICAL TRIAL: NCT07345754
Title: Women Supporting Women Using Local Solutions to Improve Infant and Young Child Feeding and Care Practices in Punjab, Pakistan
Brief Title: Women Supporting Women to Improve Infant and Child Feeding Practices in Pakistan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Rosemin Kassam, Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H21-02085
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Malnutrition in Children
Keywords: 28-day behaviour change program; Positive Deviance Hearth; Malnutrition; Feeding parctices; Pakistan
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Intervention Model Description: In Rahim Yar Khan, three union councils (UCs) were selected for the intervention arm, and three UCs were assigned to the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention arm will participate in a 28-day behaviour change program consisting of two-week cycles of Hearth sessions followed by two weeks of home visits to reinforce and practise the newly learned behaviours. Before starting the program, each index child will be referred to a local health clinic for a medical assessment and confirmation of immunization. They will receive vitamin A supplementation and deworming treatment in accordance with national protocol, if required. The intervention arm will undergo the same evaluations as the control arm, including baseline and 6-month follow-up surveys, as well as monthly anthropometric measurements.
  Interventions: Behavioral: 28-day Behavioural Change Program
- Control arm (No Intervention): This arm will not participate in the 28-day behaviour change program and will not not undergo a health facility-based assessment at baseline. The evaluations for this arm will include baseline and follow-up surveys, and monthly anthropometric measurements for up to 6 months. This group will continue to receive routine care from lady health workers (LHWs) and access health services as usual.

INTERVENTIONS:
Behavioral: 28-day Behavioural Change Program — The study's intervention includes a 28-day program with group sessions in a home-like setting (Hearth) where mothers of moderately malnourished children and family members learn practical ways to prepare nutritious meals and improve caregiving practices. Each cycle has two parts:
  Group Hearth Sessions (2 weeks): About 15 mother-child pairs attend sessions. Sessions will focus on knowledge about complementary feeding, active feeding, hygiene, caregiving, and health-seeking behaviours. Mothers will take part in cooking and caring demonstrations, rotating through roles to build hands-on skills.
  Home Practice (2 weeks): Field staff visit each home three times per week to reinforce new behaviours, provide guidance, and monitor progress.
  Mothers contribute small items such as eggs, rice, or utensils to reflect real-life conditions, while the project provides pots, utensils, and most of the food. This shared approach promotes engagement and helps sustain improved practices at home.
  Arms: Intervention arm

SUMMARY:
This project aims to reduce child malnutrition in Pakistan by building on local strengths and practical community solutions. The project focuses on children 7-23 months of age. The investigators will aim to recruit young children between 7-15 months of age, giving the youngest children priority over older children so that participants may be followed longitudinally over 6 and 12 months. The project supports participants for six months through learning, practice, and regular follow-up. The work begins with community sensitization events, where local families learn about healthy feeding for young children through group discussions, visuals, and printed materials. These sessions build awareness, encourage community support, and prepare families for the main intervention.

The core of the project is a 28-day behaviour change program. In the first two weeks, mothers and children take part in daily "Hearth" sessions, which are interactive, home-like meetings that teach practical feeding, hygiene, and caregiving skills using local foods. In the next two weeks, mothers apply learned skills at home while being visited regularly by project staff, who provide support and monitor child growth. If children gain at least 400 grams, as recommended by WHO, families graduate to monthly check-ins; if not, families may repeat the 28-day cycle up to three times. This approach targets chronic malnutrition by supporting families in adopting sustainable caregiving practices rather than providing short-term aid.

Educational materials developed with community input support the learning process. Designed with visuals and minimal text, the materials are accessible to both literate and illiterate parents and are distributed widely to encourage shared responsibility for child health.

To measure success, the project uses surveys and growth measurements for both treatment and control groups. Surveys gather information about family demographics, feeding and hygiene behaviours, and health practices, while trained staff measure children's height and weight at regular intervals. The data will help determine whether the intervention improves children's nutritional status and caregiving practices.

Ultimately, the project seeks to empower families and communities to use local resources and knowledge to support healthier child growth. The project combines community engagement, hands-on learning, and scientific evaluation to promote lasting change in how families feed, nurture, and care for young children.

DETAILED DESCRIPTION:
This study is rooted in an asset-based approach grounded in the belief that, in every community, certain individuals demonstrate uncommon behaviours that enable solutions to prevalent and seemingly intractable problems. During the formative research phase, supported by the Community Advisory Committee (CAC), the objective was to identify strategies that are already feasible within the community of Rahim Yar Khan, Pakistan, and to amplify these strategies to the wider community during the intervention phase. The intervention comprises two major components: community sensitization and a 28-day behaviour change period.

The intervention targets households with moderately malnourished children between 7 and 15 months of age and will follow and support these households for a period of six months. Consent will be obtained from both parents via thumbprint or signature. Severely malnourished children, regardless of study arm, will be referred to local health facilities for appropriate care. Households in the control group will continue with usual feeding and caregiving practices.

COMMUNITY SENSITIZATION OVERVIEW

Community sensitization events will be held in each intervention cluster. These events will introduce the project to local families and provide information on complementary feeding for children aged 6-23 months. Sessions will be delivered using a town-hall format with small group activities. Key messages, supported by visuals and printed materials from the 28-day behaviour change program (described below), will be shared with the broader community. The objective of the community sensitization component is to raise awareness about the project, disseminate best practices related to complementary feeding, and promote community buy-in, as well as neighbourhood support for households participating in the 28-day behaviour change program.

28-DAY BEHAVIOUR CHANGE PRACTICE PROGRAM OVERVIEW

Prior to recruitment and initiation of the 28-day behaviour change program, each child will undergo a health check by a physician at a local health facility. This assessment will include anemia screening and verification that all required immunizations are up to date.

The 28-day behaviour change practice includes two sequential components. The first component consists of bringing mothers and their moderately malnourished children together in a home-like setting (the Hearth) for a two-week period to rehabilitate children and promote improved feeding, hygiene, and caregiving practices. Hearth sessions will be delivered over 14 days (six Hearth days plus one rest day per week), with each session lasting approximately 2.5 hours.

The second component consists of mothers practicing the learned behaviours at home for an additional two weeks, with regular support from study staff. The Hearth and follow-up home visit model is based on the work of World Vision, which has demonstrated that behaviour change-particularly in feeding, caregiving, nurturing, and hygiene practices-may require up to three cycles for full adoption and for children to regain normal growth patterns. Accordingly, children who do not reach growth milestones after the first 28-day cycle will be offered participation in up to three cycles of the program, with non-responders referred for medical evaluation. This duration is considered optimal to minimize dependency on external rehabilitation while allowing caregivers to engage in experiential learning and subsequent practice within the household. Sessions will be facilitated by trained staff and will emphasize practical learning, including meal preparation using locally available foods.

Not all households will require three cycles. Households in which children achieve the desired weight gain of at least 400 grams, as recommended by WHO guidelines, may graduate earlier. This model is not intended to treat acute malnutrition or wasting but rather to address chronic malnutrition resulting from inadequate feeding and caregiving practices, which requires sustained engagement to reverse.

Following the Hearth sessions, mothers will continue with a 14-day at-home practice period during which newly learned behaviours are applied within the household. Study staff will visit each household three times per week for approximately 1.5 hours per visit to reinforce behaviours, monitor child growth, and provide ongoing support.

If, after each 28-day cycle, a child meets growth milestones, home visits will transition to monthly check-ins for up to six months. If growth milestones are not met, households will be invited to repeat the 28-day Hearth and home practice cycles up to three times.

To reinforce the intervention, supplemental printed materials will be distributed to households during the 28-day program. These materials will be developed in collaboration with the CAC and informed by findings from the formative research phase. Designed to be accessible to illiterate populations, the materials will feature culturally relevant visuals with minimal text and will be tailored for both men and women. An estimated 5,000 copies will be produced for dissemination to households participating in both the 28-day behaviour change program and the community sensitization activities.

EVALUATION

The project will evaluate the effectiveness of the intervention using tools adapted from existing validated instruments. These tools were informed by the formative research phase, reviewed by the CAC for clarity and cultural appropriateness, and pilot tested. All instruments have been translated into the local Punjabi dialect spoken by both Punjabi and Saraiki tribes residing in Rahim Yar Khan. Households in both the treatment and control arms will undergo similar evaluation procedures.

The evaluation will involve two primary data collection strategies.

1. BASELINE AND FOLLOW-UP SURVEYS

   Interview-assisted surveys will be conducted with mothers to collect information on demographics, child health status, infant and young child feeding (IYCF) practices, hygiene behaviours, healthcare-seeking behaviours, gender norms, psychosocial factors, and available resources. Baseline surveys will be administered after informed consent is obtained. Follow-up (endline) surveys will be conducted six months after baseline. With the exception of demographic information, which will be collected only at baseline, both baseline and endline surveys will collect the same information. A third survey at 12 months post-intervention will be conducted if funding permits.
2. ANTHROPOMETRIC MEASUREMENTS (WEIGHT AND HEIGHT)

Anthropometric data will be collected by trained study staff to measure children's height and weight using calibrated instruments to minimize observer bias. Measurements will be analyzed using WHO Anthro software to determine nutritional status based on standard Z-scores (weight-for-age, height-for-age, and weight-for-height). Children will be classified as underweight, stunted, wasted, or well-nourished. For children in both the treatment and control arms, anthropometric measurements will be collected at recruitment (as part of the baseline survey), during monthly follow-up visits, and at endline. In addition, for children in the treatment arm, weight measurements will be collected during the 28-day behaviour change practice program on Days 1, 13, and 28.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must meet all of the following conditions:

Child-Level Criteria:

While children in the intervention phase will range from ages 7-23 months, At the time of recruitment children will range from Ages: 7-15 months.

* Priority will be given to younger children, aged 7-11 months, followed by 12-15 months to allow completion of the intervention and follow-up visits before the child turns 24 months of age, as complementary feeding refers to feeding practices between the ages of 6-24 months.
* Moderate malnutrition, defined by: Weight-for-age Z-score between -2 and -3 standard deviations.

Household-Level Criteria:

Households will be eligible to participate if:

* They meet the classification of very poor or poor (based on community-defined wealth stratification).
* Have access to clean water and sanitation.
* Food secure at time of recruitment, defined as:

  * On government assistant program or at least one adult has permanent employment, or two or more have temporary employment.
  * Ownership of at least one simple livestock (e.g., chicken, goat, or sheep) or express willingness to accept and care for livestock provided by the project team.
  * Access to a kitchen garden, or willingness to establish one with study support

Mother Eligibility Criteria:

The household is eligible only if the mother meets all of the following:

1. Mother is the primary caregiver for the Index Child (responsible for daily care, including supervision, bathing, and feeding).
2. Mother is alive and at least 18 years old.
3. Mother is currently breastfeeding the Index Child and willing to continue until the child reaches 2 years of age.
4. Mother expresses an interest in participating in the PD/Hearth program.
5. Mother agrees to attend up to three Hearth sessions.
6. Mother is willing and able to contribute to one of the following for Hearth sessions:

   * "Special" food items (e.g., apple, banana, carrot, chickpea, egg, garlic, lentils, rice, spinach, tomato, etc.), or
   * Other essential items (e.g., utensils, bowls, spoons, soap, nail cutter, towels, water, mat, salt, matchstick).
7. Mother provides permission for study follow-ups as outlined above.
8. Mother agrees to a full medical check-up for the Index Child at the nearest public health facility, including a one-time hematocrit finger-prick test (Hb test).
9. Mother provides informed consent via thumbprint or written signature.

Exclusion Criteria:

Child-Level Exclusions:

* Children who are Severely malnourished, mildly underweight or of normal weight.
* Children with Physical disabilities: difficulty in seeing, hearing, picking up small objects with his/her hand.
* Children with chronic illnesses that may interfere with normal growth (based on past or current medical history):
* Malabsorption
* Chronic Kidney Disease
* Inflammatory Bowel Disease
* Congenital Heart Disease
* Endocrine Disorders (e.g., hypothyroidism, growth hormone deficiencies)
* Chronic Respiratory Diseases (e.g., asthma, lung diseases)
* Congenital or Acquired Immunodeficiency, and Neurological Disorders

Household-Level Exclusion:

• Households who do not meet the inclusion criteria.

Ages: 7 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight | At baseline; Hearth Days 1, 13, 28; During monthly home visits; End-Survey after 6 months
  Index Child's weight will be measured in Kilogram(Kg) and will be used to assess the Index child's nutritional status.
Weight-for-age Z-score | At baseline; Hearth Days 1, 13, 28; During monthly home visits; End-Survey after 6 months
  Nutritional status of Index child will classify as (1) severely underweight, (2) moderate underweight, (3) mild underweight, (4) well-nourished or normal weight using weight-for-age Z-score as below.
  Severely underweight if weight-for-age Z-score <-3 SD of the median. Moderate underweight if weight-for-age Z-score between -2 SD and -3 SD. Mild underweight if weight-for-age Z-score between -1 SD and -2 SD. Normal weight if weight-for-age Z-score between -1 SD and +1 SD.

SECONDARY OUTCOMES:
Length | At baseline and 6 months post-intervention
  Index Child's length will be measured in centimeters(cm) and will be used to assess the Index child's nutritional status and Height-for-Age Z-score.
Height-for-age Z-score | At baseline and 6 months post-intervention
  Length measurement will be used to classify Index child as (1) severely stunted, (2) moderately stunted, (3) mildly stunted, (4) Normal length using length/height-for-age Z-score.
  Severe stunting if length/height-for-age Z-score <-3 SD of the median. Moderate stunting if length/height-for-age Z-score between -2 SD and -3 SD. Mild stunting if length/height-for-age Z-score between -1 SD and -2 SD. Normal length if length/height-for-age Z-score between -1 SD and +1 SD.
Mid-upper arm circumference (MUAC) | At baseline and 6 months post-intervention
  MUAC measurement for Index child will be assessed to classify (1) Green >12.5 cm, (2) Yellow 11.5-12.5 cm and (3) Red <11.5 cm.
Weight-for-Height Z-Score | At baseline and 6 months post-intervention
  This measurement assesses how the child's weight compares to the median weight of children their same age and height. Sign of wasting classify as (1) severe wasting, (2) moderate wasting, (3) marginal wasting, (4) well-nourished
MINIMUM MEAL FREQUENCY 6-23 MONTHS (MMF) | At baseline and 6 months post-intervention
  Percentage of children 6-23 months of age who consumed solid, semi-solid or soft foods (but also including milk feeds for non-breastfed children) the minimum number of times or more during the previous day.
  This indicator is measured using the "24-hr food recall questionnaire" on the baseline and 6-month follow-up surveys.
  Numerator:
  Breastfed children 6-23 months of age who consumed solid, semi-solid or soft foods the minimum number of times or more during the previous day; OR Non-breastfed children 6-23 months of age who consumed at least four solid, semi-solid or soft food feeds or milk feeds during the previous day, with at least one of the four being a solid, semi-solid or soft food feed.
  Denominator: Children 6-23 months of age.
MINIMUM DIETARY DIVERSITY 6-23 MONTHS (MDD) | At baseline and 6 months post-intervention
  Percentage of children 6-23 months of age who consumed solid, semi-solid or soft foods (but also including milk feeds for non-breastfed children) the minimum number of times or more during the previous day.
  This indicator will be assessed using the "24-hr food recall questionnaire" on the baseline and 6-month follow-up surveys.
  Numerator:
  Breastfed children 6-23 months of age who consumed solid, semi-solid or soft foods the minimum number of times or more during the previous day; OR Non-breastfed children 6-23 months of age who consumed at least four solid, semi-solid or soft food feeds or milk feeds during the previous day, with at least one of the four being a solid, semi-solid or soft food feed.
  Denominator:
  Children 6-23 months of age.

CONTACTS AND LOCATIONS:
Locations (1):
- RYK, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-10-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT07345754/Prot_000.pdf